CLINICAL TRIAL: NCT07371663
Title: An Open-Label, Multicenter Phase Ib/II Clinical Trial of TCC1727 in Combination With Benmelstobart/Olaparib/Topotecan for Advanced Solid Tumors
Brief Title: An Phase Ib/II Clinical Trial of TCC1727 Combination Therapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCC1727-II-01
Record Dates: First submitted 2025-12-15; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Solid Cancers; NSCLC (Advanced Non-small Cell Lung Cancer); Gastric (Stomach) Cancer; Endometrial Cancer; Malignant Melanoma
Keywords: Ataxia Telangiectasia and Rad3-related protein inhibitor; Advanced solid tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Endometrial Neoplasms; Melanoma; Ataxia Telangiectasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TCC1727 + benmelstobart (Dose Level 1) (Experimental): TCC1727 tablets 90 mg orally twice daily (bid) in 21-day cycles combined with benmelstobart injection 1200 mg by intravenous infusion in 21-day cycles until disease progression
  Interventions: Drug: TCC1727 tablet 90mg; Combination Product: benmelstobart Injection
- TCC1727 + benmelstobart (Dose Level 2) (Experimental): TCC1727 tablets 120 mg orally twice daily (bid) in 21-day cycles combined with benmelstobart injection 1200 mg by intravenous infusion in 21-day cycles until disease progression
  Interventions: Drug: TCC1727 tablet 120mg; Combination Product: benmelstobart Injection
- TCC1727 + benmelstobart (Dose Level 3) (Experimental): TCC1727 tablets 160 mg orally twice daily (bid) in 21-day cycles combined with benmelstobart injection 1200 mg by intravenous infusion in 21-day cycles until disease progression
  Interventions: Drug: TCC1727 tablet 160mg; Combination Product: benmelstobart Injection

INTERVENTIONS:
Drug: TCC1727 tablet 90mg — TCC1727 tablets 90 mg, orally, twice daily (bid), continuous dosing in 21-day cycles until disease progression
  Arms: TCC1727 + benmelstobart (Dose Level 1)
Drug: TCC1727 tablet 120mg — TCC1727 tablets 120 mg, orally, twice daily (bid), continuous dosing in 21-day cycles until disease progression
  Arms: TCC1727 + benmelstobart (Dose Level 2)
Drug: TCC1727 tablet 160mg — TCC1727 tablets 160 mg, orally, twice daily (bid), continuous dosing in 21-day cycles until disease progression
  Arms: TCC1727 + benmelstobart (Dose Level 3)
Combination Product: benmelstobart Injection — Administer 1200 mg per dose via intravenous infusion on Day 1 of every 3-week cycle until disease progression.

SUMMARY:
This is a Phase Ib/II clinical study. The Phase Ib dose-escalation study aims to evaluate and determine the recommended Phase II dose (RP2D) of TCC1727 in combination with benmelstobart /olaparib /topotecanfor patients with advanced solid tumors.

The Phase II expansion study will assess the efficacy and safety of TCC1727 combined with benmelstobart /olaparib/topotecanin selected advanced solid tumor indications.

The study pre-specifies three treatment combinations, with Combination 1 (TCC1727 + benmelstobart) being prioritized for initial evaluation. The decision to proceed with Combination 2 and Combination 3will be based on clinical data from Combination 1.

ELIGIBILITY:
Inclusion Criteria:

* -Voluntarily participate in this study and sign the informed consent form.
* At the time of signing the informed consent, subjects must be ≥18 years of age (inclusive).
* Subjects must have histologically or cytologically confirmed advanced or metastatic solid tumors and have experienced disease progression following prior standard anti-tumor therapy; or subjects must have no available standard therapy, be intolerant to or refuse standard therapy, or meet the specific requirements for the corresponding phase and group as follows:

  * Phase Ib :Subjects with advanced, recurrent, or refractory solid tumors, which may include (but are not limited to) the specific tumor types in Phase II.
  * Phase II Study:Based on different combination therapy groups, subjects with the following specific tumor types (different population cohorts):

TCC1727 combined with Benmelstobart Group:

The study will enroll subjects with advanced solid tumors lacking standard therapies, including but not limited to non-small cell lung cancer (NSCLC), endometrial cancer, and other advanced solid tumors (e.g., colorectal cancer, urothelial carcinoma, gastric cancer, and gastroesophageal junction cancer):

Cohort 1 (NSCLC):Patients with histologically or cytologically confirmed locally advanced or metastatic NSCLC who are eligible for second- or third-line therapy. Patients must have received prior therapy with an anti-PD-(L)1-containing regimen (either as monotherapy or in combination) and a platinum-based doublet regimen for locally advanced or metastatic NSCLC.

Subgroup 1: ATM mutation. Subgroup 2: ATM wild-type, with or without other DDR functional defects.

Cohort 2 (Endometrial Cancer):Patients with histopathologically confirmed recurrent or metastatic advanced endometrial cancer who have received at least one prior platinum-based chemotherapy and immune checkpoint inhibitor (PD-1 or PD-L1) therapy (sequential or concurrent therapy allowed; sequential therapy refers to platinum-based chemotherapy followed by immune checkpoint inhibitor maintenance therapy).

Subgroup 1: DDR functional defect, ATM wild-type or mutated. Subgroup 2: DDR functional normal.

Cohort 3 (Other Advanced Solid Tumors):Patients with histologically or cytologically confirmed advanced malignant solid tumors who have failed standard therapy, are intolerant to standard therapy, have no standard therapy available, or for whom standard therapy is currently unsuitable.

Subgroup 1: DDR functional defect, ATM wild-type or mutated. Subgroup 2: DDR functional normal.

TCC1727 combined with Olaparib Tablets Group:

The study will enroll subjects with histopathologically confirmed recurrent ovarian cancer:

Cohort 4 (Ovarian Cancer):Subjects with histopathologically confirmed recurrent epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer:

Subgroup 1: Subjects who have experienced disease progression after prior Olaparib Tablets therapy (maintenance or subsequent therapy). Subjects must not have received further treatment after progression on Olaparib Tablets.

Subgroup 2: Subjects who have not received Olaparib Tablets and have primary platinum-resistant/refractory disease (recurrence within 6 months of last platinum-based therapy). Subjects must have received ≤3 prior lines of therapy since developing platinum resistance.

TCC1727 combined with Topotecan Hydrochloride for Injection Group:

The study will enroll subjects with histopathologically or cytologically confirmed small cell lung cancer (SCLC):

Cohort 5 (SCLC):Subjects who have progressed after platinum-based chemotherapy combined with PD-(L)1 therapy, or subjects with extensive-stage SCLC who have relapsed or progressed within ≤6 months after first-line therapy.

* At least one measurable lesion (per RECIST v1.1; lesions previously treated with local therapy may be considered target lesions if they show clear progression per RECIST v1.1).
* Subjects must provide sufficient tumor tissue samples, including but not limited to fresh specimens (preferred) or formalin-fixed, paraffin-embedded (FFPE) tumor tissue obtained within approximately 24 months prior to randomization, unstained FFPE slides, or core needle biopsy tissue for biomarker testing.
* ECOG performance status score of 0-1 within 7 days prior to the first dose of study drug.
* Expected survival ≥12 weeks.
* Ability to swallow tablets whole and maintain this method of administration.
* Organ function within the following ranges within 7 days prior to the first dose of study drug (no blood component or growth factor therapy within 14 days prior to the first dose):

  1. Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L;
  2. White blood cell count (WBC) ≥3.0 × 10⁹/L;
  3. Platelet count ≥100 × 10⁹/L;
  4. Hemoglobin (Hb) ≥90 g/L;
  5. Serum albumin ≥30 g/L;
  6. Total bilirubin ≤1.5 × ULN (≤2.0 × ULN for hepatocellular carcinoma or subjects with liver metastases);
  7. ALT and AST ≤3 × ULN (≤5.0 × ULN for hepatocellular carcinoma or subjects with liver metastases);
  8. Alkaline phosphatase (ALP) ≤2.5 × ULN (≤5 × ULN if bone metastases are present);
  9. Serum creatinine ≤1.5 × ULN or creatinine clearance (CrCL) ≥60 mL/min (Cockcroft-Gault formula);
  10. APTT ≤1.5 × ULN and INR or PT ≤1.5 × ULN (for subjects not receiving anticoagulation therapy);
  11. QTc <450 ms (male) or <470 ms (female), LVEF ≥50%.
* For non-sterilized or fertile female subjects, medically approved contraception (e.g., intrauterine device, oral contraceptives, or condoms) must be used during the study and for 6 months after the last dose. Non-sterilized female subjects must have a negative serum HCG test within 72 hours before the first dose and must not be breastfeeding. Male subjects with fertile partners must use effective contraception during the study and for 3 months after the last dose.

Exclusion Criteria:

* Known primary central nervous system (CNS) tumors (including meningeal tumors); symptomatic brain metastases, spinal cord compression, carcinomatous meningitis, or uncontrolled CNS metastases. Exceptions: Subjects with completely resected and/or irradiated CNS metastases that are stable or improved for ≥4 weeks before screening (no evidence of brain edema and no need for corticosteroids or anticonvulsants). Asymptomatic brain metastases <1 cm in diameter without surrounding edema are also allowed.
* Major surgery, radiotherapy, chemotherapy, or other investigational anti-tumor therapy completed <4 weeks before the first dose (exceptions: small-molecule anti-tumor therapy completed >5 half-lives or >10 days before the first dose, whichever is longer; palliative radiotherapy completed >2 weeks before the first dose).
* Use of strong CYP3A4 inhibitors or inducers within 14 days before the first dose (e.g., rifampin, rifapentine, St. John's wort, carbamazepine, phenytoin, barbiturates, ketoconazole, itraconazole, clarithromycin, voriconazole, atazanavir, ritonavir, saquinavir, grapefruit juice).
* Any unresolved ≥Grade 2 toxicity (per CTCAE v5.0) from prior anti-tumor therapy (except alopecia, pigmentation, or laboratory abnormalities meeting inclusion criteria).
* Inability to swallow tablets, gastrointestinal dysfunction, or any condition that may affect drug absorption (per investigator's judgment).
* Uncontrolled severe diseases, including:

  1. Poorly controlled hypertension (systolic BP ≥150 mmHg or diastolic BP ≥100 mmHg);
  2. Clinically significant cardiovascular disease within 6 months before the first dose (e.g., myocardial infarction, severe/unstable angina, stroke, ≥Grade 2 congestive heart failure [NYHA classification]);
  3. Arrhythmia (≥Grade 2 per CTCAE v5.0, including QTcF ≥450 ms [male] or ≥470 ms [female]);
  4. Unexplained fever ≥38.5°C within 14 days before the first dose or active infection requiring systemic therapy;
  5. Active viral hepatitis (HBV DNA ≥500 IU/mL for HBsAg-positive and/or anti-HBc-positive subjects; HCV RNA-positive for anti-HCV-positive subjects; antiviral therapy required for eligible HBV/HCV-positive subjects);
  6. Active syphilis;
  7. Active tuberculosis;
  8. Immunodeficiency (e.g., HIV-positive, congenital/acquired immunodeficiency, organ transplant history);
  9. Poorly controlled diabetes (fasting blood glucose >10 mmol/L).
* Uncontrolled pleural effusion, pericardial effusion, ascites, or recurrent ascites requiring drainage within 28 days before the first dose.
* Significant bleeding symptoms or tendency within 3 months before the first dose.
* Chronic systemic corticosteroid therapy (>10 mg prednisone equivalent daily) or immunosuppressive therapy within 14 days before the first dose.
* Active autoimmune disease requiring systemic treatment within the past 2 years (e.g., immunomodulators, corticosteroids, immunosuppressants). Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement for adrenal/pituitary insufficiency) is allowed. (Applies only to Ib Phase and Phase II TCC1727 + Benmelstobart groups.)
* History of severe allergic reactions to study drugs or their excipients.
* Other malignancies within 3 years before screening (except cured basal cell carcinoma, cervical carcinoma in situ, or thyroid papillary carcinoma).
* Prior ≥Grade 3 immune-mediated adverse events (imAEs) or permanent discontinuation due to imAEs during anti-PD-(L)1 therapy.
* Prior treatment with TCC1727, other ATR inhibitors, or cell cycle checkpoint inhibitors (e.g., ATM inhibitors, WEE1 inhibitors, CHK1/CHK2 inhibitors).
* Other severe physical/mental illnesses or factors that may increase study risk or interfere with results, or any condition deemed unsuitable by the investigator.

Additional exclusions:

* Phase II Cohort 1 (NSCLC):Exclude subjects with known EGFR, ALK, ROS1, BRAF, MET, RET, or RAS mutations; exclude mixed NSCLC/SCLC histology.
* Phase II Cohort 2 (Endometrial Cancer):Exclude uterine carcinosarcoma, endometrial leiomyosarcoma, or endometrial stromal sarcoma.
* Phase II Cohort 3 (Other Solid Tumors):Exclude KRAS/NRAS/BRAF mutations or MSI-H status.
* Phase II Cohort 4 (Ovarian Cancer) & Ib Phase TCC1727 + Olaparib Tablets: Exclude prior myelodysplastic syndrome or acute myeloid leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib：To determine dose-limiting toxicity (DLT) at each dose level | 21 Days
  Dose Escalation To observe the tolerability and safety of TCC1727 combination therapy.
MTD | 21 days
  The maximum tolerated dose (MTD) of TCC1727 in combination with benmelstobart/olaparib/topotecan will be determined based on safety, tolerability, kinetics, preliminary efficacy, and other available data
RP2D | 21 days
  The recommended Phase II dose (RP2D) of TCC1727 in combination with benmelstobart/olaparib/topotecan will be determined based on safety, tolerability, kinetics, preliminary efficacy, and other available data
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 21days
  Adverse events (AEs) were assessed according to NCI-CTCAE v5.0, including severity grading of abnormal findings in laboratory tests, vital signs, physical examinations, and electrocardiograms (ECGs) from signing of informed consent through the end of the safety follow-up period or prior to the start of a new anticancer therapy

SECONDARY OUTCOMES:
Assess objective response rate (ORR: complete response + partial response), based on RECIST 1.1 | 6 month
  Efficacy evaluation was performed every 6 weeks (± 7 days), extended to 9 weeks (± 7 days) after 8 cycles for efficacy evaluation, and patients were assessed for tumor by the investigator according to RECIST v1.1
PK parameters of TCC1727 | Day1, Day22
  Blood samples were collected before and after administration of C1, C2 to evaluate the kinetic (PK) parameters of TCC1727: Cmax
PK parameters of TCC1727 | Day1, Day22
  Blood samples were collected before and after administration of C1, C2 to evaluate the kinetic (PK) parameters of TCC1727: Tmax
PK parameters of TCC1727 | Day1, Day22
  Blood samples were collected before and after administration of C1, C2 to evaluate the kinetic (PK) parameters of TCC1727: Trough concentration (minimum concentration at steady state)-Ctrough
AUC0-t | Day1, Day22
  Blood samples were collected before and after administration of C1, C2 to evaluate the kinetic (PK) parameters of TCC1727:AUC0-t
AUC0-∞ | Day1, Day22
  Blood samples were collected before and after administration of C1, C2 to evaluate the kinetic (PK) parameters of TCC1727:AUC0-∞
PK parameters of TCC1727 | Day1, Day22
  Blood samples were collected before and after administration of C1, C2 to evaluate the kinetic (PK) parameters of TCC1727:t1/2
PK parameters of TCC1727 | Day1, Day22
  Blood samples were collected before and after administration of C1, C2 to evaluate the kinetic (PK) parameters of TCC1727:Clearance
PK parameters of TCC1727 | Day1, Day22
  Blood samples were collected before and after administration of C1, C2 to evaluate the kinetic (PK) parameters of TCC1727:Volume of distribution at steady state （Vss）
Assess disease control rate (DCR) based on RECIST 1.1; | 6 month
  Efficacy evaluation was performed every 6 weeks (± 7 days), extended to 9 weeks (± 7 days) after 8 cycles for efficacy evaluation, and patients were assessed for tumor by the investigator according to RECIST v1.1
Assess duration of response (DoR) based on RECIST 1.1 | 6 month
  Efficacy evaluation was performed every 6 weeks (± 7 days), extended to 9 weeks (± 7 days) after 8 cycles for efficacy evaluation, and patients were assessed for tumor by the investigator according to RECIST v1.1
Assess time to response (TTR) based on RECIST 1.1 | 6 month
  Efficacy evaluation was performed every 6 weeks (± 7 days), extended to 9 weeks (± 7 days) after 8 cycles for efficacy evaluation, and patients were assessed for tumor by the investigator according to RECIST v1.1
Assess progression-free survival (PFS) based on RECIST 1.1 | 6 month
  Efficacy evaluation was performed every 6 weeks (± 7 days), extended to 9 weeks (± 7 days) after 8 cycles for efficacy evaluation, and patients were assessed for tumor by the investigator according to RECIST v1.1
Assess overall survival (OS) of subjects | 12 month
  Survival follow-up assessments will be conducted at 12-week intervals (±7 days) to document Overall survival(OS) and subsequent anticancer therapies, with follow-up terminating at the earliest occurrence of study completion, death, loss to follow-up, or patient withdrawal

OTHER OUTCOMES:
Baseline tumor tissue predictive biomarkers | Screening visit（Day-28 to Day1）
  including but not limited to the correlation between PD-L1 expression, tumor mutational burden (TMB)-related gene mutation status, and the efficacy of TCC1727 combined with benmelstobart in subjects with advanced solid tumors
Correlation between mutation status of DDR-related genes in baseline tumor tissues and efficacy of TCC1727 combination therapy | Screening visit（Day-28 to Day1）
  Mutation status of DDR-related genes in baseline tumor tissue including but not limited to correlation of ATM mutations with efficacy of TCC1727 in combination with Benmelstobart/olaparib/topotecan in subjects with advanced solid tumors
Before and after treatment, the distribution changes of blood immune cells . (only applicable to the combination with Benmelstobart) | Screening visit（Day-28 to Day1）, Cycle1Day8, Cycle1Day15, Cycle2Day1(Each cycle is 21days)
  The changes in the distribution of blood immune cells at screening period and Cycle1D8, Cycle1D15 and Cycle2D1 . (only applicable to the combination with Benmelstobart)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided